CLINICAL TRIAL: NCT04229368
Title: Effect of Vitamin D Status and Repletion on Postoperative Total Joint Arthroplasty Complications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); Newton-Wellesley Hospital (Other)
Responsible Party: Principal Investigator, Antonia Faustina Chen, Director of Research Arthroplasty Division, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2018P001701
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Hip Arthropathy; Knee Arthropathy; Vitamin D Deficiency
Keywords: joint replacement; hip arthroplasty; knee arthroplasty; clinical outcomes; Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Prospective randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 900 patients to be enrolled total including controls, and two additional study arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Vitamin D3 Supplementation (Active Comparator): Subjects enrolled into Group 1 (low-dose Vitamin D3 supplementation) will receive 800 IU of oral Vitamin D3 (Cholecalciferol) daily for 4 weeks prior to surgery, followed by 800 IU of oral Vitamin D3 daily for 3 months after surgery. Vitamin D3 supplementation will be given for a total of 4 months. Supplementing Vitamin D-deficient patients with a minimum of 800 IU of Vitamin D3 daily is supported by the IOM.
  Interventions: Dietary Supplement: Vitamin D3
- High Vitamin D3 Supplementation (Active Comparator): Subjects enrolled into Group 2 (high-dose Vitamin D3 supplementation) will receive 50,000 IU of oral Vitamin D3 (Cholecalciferol) twice per week for 1 weeks followed by 50,000 IU once per week for 3 weeks prior to surgery. After surgery they will receive 50,000 IU of oral Vitamin D3 once per week for 4 weeks followed by 800 IU daily for 8 weeks. Vitamin D3 supplementation will be given for a total of 4 months.
  Interventions: Dietary Supplement: Vitamin D3
- No supplementation (No Intervention): Subjects with serum 25(OH)D level ≥30ng/mL will not receive any Vitamin D supplementation both pre- and postoperatively, as these are considered sufficient. These control patients will be asked to take any supplements containing Vitamin D for the duration of their participation in the trial. All patients in group 3 will have their serum 25(OH)D checked at 3 months after the surgery.

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Vitamin D will be given at doses commonly given to patients with low vitamin D levels
  Other Names: cholecalciferol
  Arms: High Vitamin D3 Supplementation; Low Vitamin D3 Supplementation

SUMMARY:
Vitamin D status has been shown to have an effect on post-operative outcomes in total joint arthroplasty. The goal of this study is to determine if pre-operative supplementation and correction of Vitamin D deficiency can reduce postoperative complications.

DETAILED DESCRIPTION:
Total joint arthroplasty (TJA) is one of the most common surgical procedures performed in the United States (US), with approximately 2.5 million individuals with total hip arthroplasties (THAs) and 4.7 million individuals with total knee arthroplasties (TKAs) in 2010. Patients who undergo TJA commonly have Vitamin D deficiency, with rates reported to be 24-61% in primary TJA patients. Vitamin D deficiency affects women and minorities at high rates, in addition to non-Hispanic whites. Previous studies demonstrated that Vitamin D deficiency poorly impacts outcomes after various surgical procedures. Specifically in TJA patients, recent studies show a higher rate of Vitamin D deficiency in periprosthetic joint infection (PJI) patients, and a higher rate of postoperative complications and infection in revision TJA patients with low Vitamin D. In a PJI mouse model, Vitamin D-deficient mice were shown to have an increased bacterial burden when compared to Vitamin D-deficient mice that received "rescue" cholecalciferol (Vitamin D3) supplementation. Bacterial burden was similarly decreased between normal mice and the Vitamin D-deficient "rescue" mice receiving supplementation. A single dose of Vitamin D3 supplementation in Vitamin D-deficient mice using the same mouse model reversed the effect of PJI by decreasing bacterial burden and neutrophil infiltration.

The serum concentration of 25-hydroxycholecalciferol or 25-hydroxyvitamin D (25(OH)D) is the most accurate measure of stores of Vitamin D in the body. There are currently different recommendations regarding the optimal serum 25(OH)D level for bone health, the optimal daily intake of Vitamin D, and the treatments for Vitamin D deficiency or insufficiency. These controversial topics do not provide clear clinical guidance on how to optimize Vitamin D levels in surgical patients to reduce complication rates. The US Institute of Medicine (IOM) committee recommended a 25(OH)D level >20 ng/mL but other organizations recommend ≥30 ng/mL. At present, deficient levels of Vitamin D are generally defined as a 25(OH)D <20 ng/ml, relative insufficiency as 20 to 29 ng/mL, and sufficient levels as ≥ 30 ng/ml. In 2011, the IOM established Recommended Dietary Allowances (RDAs) for Vitamin D of 600-800 IU/d in order to achieve a 25(OH)D level of 20 ng/ml for 97.5% of the general population. The debate concerns recommendations based upon population science, in contrast to care of an individual patient. Thus, there is continuing debate among several groups that recommend higher Vitamin D3 doses and 25(OH)D levels of ≥30 ng/mL for optimal bone health and in high-risk individuals with osteoporosis. The National Osteoporosis Foundation recommends 800 to 1000 IU Vitamin D3 daily for adults aged 50 years and older, as do the International Osteoporosis Foundation and Endocrine Society. The Endocrine Society recommended even higher doses up to 1500 to 2000 IU/d of Vitamin D3 for older adults. For Vitamin D deficiency, the recommended treatment is 50,000 units of Vitamin D3 weekly for 8 weeks with an assay repeat to determine whether Vitamin D-sufficiency ≥30ng/mL was achieved. The proposed study was designed in light of debated recommendations in the literature and should result in rigorous new information about 25(OH)D levels achieved with different doses of Vitamin D3 supplementation and their impact on post-TJA complications.

There are no current studies in literature examining whether preoperative supplementation and correction of Vitamin D deficiency may reduce complications following TJA. The aim of this randomized controlled trial is to evaluate the ability of different doses (low and high dose) of Vitamin D3 supplementation to affect adverse events and functional outcomes following total joint arthroplasty surgery. To conduct this study, investigators propose randomizing subjects with 25(OH)D levels between 10 and 29 ng/mL to receive different doses of Vitamin D to assess the effects of Vitamin D3 supplementation dosage on postoperative TJA complication rates. Consented patients with serum 25(OH)D levels equal or greater than 30 ng/dL will be included in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years of age undergoing elective unilateral primary TJA for osteoarthritis
* Patients with a pre-operative serum 25(OH)D levels ≥10 ng/mL
* Patients who consent to the study

Exclusion Criteria:

* Adult patients ≥18 years of age undergoing elective primary TJA with a pre-operative serum 25(OH)D2,3 level <10 ng/mL
* Patients undergoing revision surgery
* Patients lacking mental capacity to comply with study procedures
* Patients with serum 25(OH)D levels between 10-29 ng/dL refusing to stop their current Vitamin D and multivitamins supplementations
* Hypercalcemia (total calcium >10.6 mg/dL or ionized serum calcium >5.4mg/dL)
* History of nephrolithiasis
* Granulomatous disease
* Dialysis and advanced kidney disease
* Previous infection/septic arthritis
* Inability to swallow Vitamin D3 pills
* Allergy to Vitamin D3 (It is estimated that 1 in 300 individuals may have an allergy with skin manifestations 17)
* Hypocalcemia (<8.5 mg/dL)
* Chronic kidney disease (eGFR <60 mL/minute)
* Known hyperparathyroidism
* Known osteoporosis/insufficiency stress fractures (if normal stresses are applied to an abnormal bone)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Readmission, reoperation, wound complications, and PJI | Preoperative visit to three months post-op
  adverse events

SECONDARY OUTCOMES:
Vitamin D status | Day of surgery to to three months post-op
  Vitamin D levels will be drawn initially, during supplementation and following
Patient-Reported Outcomes Measurement Information System (PROMIS) | Preoperative visit to three months post-op
  set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children.41 to 78.3 with higher scores representing worse pain impact.
Pain Levels: visual analog scale (VAS) | Preoperative visit to three months post-op
  Scores on the VAS pain scale range from 0-10 with 0 being no pain and 10 being the highest pain level imaginable.
Hip disability and Osteoarthritis Outcome Score (HOOS) | Preoperative visit to three months post-op
  Scores range from 0 to 100 with a score of 0 indicating the worst possible hip symptoms and 100 indicating no hip symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Antonia F Chen, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Maradit Kremers H, Larson DR, Crowson CS, Kremers WK, Washington RE, Steiner CA, Jiranek WA, Berry DJ. Prevalence of Total Hip and Knee Replacement in the United States. J Bone Joint Surg Am. 2015 Sep 2;97(17):1386-97. doi: 10.2106/JBJS.N.01141. PMID 26333733
- [Background] Nawabi DH, Chin KF, Keen RW, Haddad FS. Vitamin D deficiency in patients with osteoarthritis undergoing total hip replacement: a cause for concern? J Bone Joint Surg Br. 2010 Apr;92(4):496-9. doi: 10.1302/0301-620X.92B3.23535. PMID 20357324
- [Background] Jansen JA, Haddad FS. High prevalence of vitamin D deficiency in elderly patients with advanced osteoarthritis scheduled for total knee replacement associated with poorer preoperative functional state. Ann R Coll Surg Engl. 2013 Nov;95(8):569-72. doi: 10.1308/rcsann.2013.95.8.569. PMID 24165338
- [Background] Forrest KY, Stuhldreher WL. Prevalence and correlates of vitamin D deficiency in US adults. Nutr Res. 2011 Jan;31(1):48-54. doi: 10.1016/j.nutres.2010.12.001. PMID 21310306
- [Background] Taksler GB, Cutler DM, Giovannucci E, Keating NL. Vitamin D deficiency in minority populations. Public Health Nutr. 2015 Feb;18(3):379-91. doi: 10.1017/S1368980014000457. Epub 2014 Apr 15. PMID 25112179
- [Background] Maier GS, Horas K, Seeger JB, Roth KE, Kurth AA, Maus U. Is there an association between periprosthetic joint infection and low vitamin D levels? Int Orthop. 2014 Jul;38(7):1499-504. doi: 10.1007/s00264-014-2338-6. Epub 2014 Apr 16. PMID 24737149
- [Background] Traven SA, Chiaramonti AM, Barfield WR, Kirkland PA, Demos HA, Schutte HD, Drew JM. Fewer Complications Following Revision Hip and Knee Arthroplasty in Patients With Normal Vitamin D Levels. J Arthroplasty. 2017 Sep;32(9S):S193-S196. doi: 10.1016/j.arth.2017.02.038. Epub 2017 Mar 8. PMID 28372917
- [Background] Iglar PJ, Hogan KJ. Vitamin D status and surgical outcomes: a systematic review. Patient Saf Surg. 2015 Apr 30;9:14. doi: 10.1186/s13037-015-0060-y. eCollection 2015. PMID 25926889
- [Background] Walker JP, Hiramoto JS, Gasper WJ, Auyang P, Conte MS, Rapp JH, Lovett DH, Owens CD. Vitamin D deficiency is associated with mortality and adverse vascular access outcomes in patients with end-stage renal disease. J Vasc Surg. 2014 Jul;60(1):176-83. doi: 10.1016/j.jvs.2014.01.037. Epub 2014 Feb 28. PMID 24582700
- [Background] Hegde V, Dworsky EM, Stavrakis AI, Loftin AH, Zoller SD, Park HY, Richman S, Johansen D, Hu Y, Taylor JA, Hamad CD, Chun RF, Xi W, Adams JS, Bernthal NM. Single-Dose, Preoperative Vitamin-D Supplementation Decreases Infection in a Mouse Model of Periprosthetic Joint Infection. J Bone Joint Surg Am. 2017 Oct 18;99(20):1737-1744. doi: 10.2106/JBJS.16.01598. PMID 29040128
- [Background] Cosman F, de Beur SJ, LeBoff MS, Lewiecki EM, Tanner B, Randall S, Lindsay R; National Osteoporosis Foundation. Clinician's Guide to Prevention and Treatment of Osteoporosis. Osteoporos Int. 2014 Oct;25(10):2359-81. doi: 10.1007/s00198-014-2794-2. Epub 2014 Aug 15. PMID 25182228
- [Background] Dawson-Hughes B, Mithal A, Bonjour JP, Boonen S, Burckhardt P, Fuleihan GE, Josse RG, Lips P, Morales-Torres J, Yoshimura N. IOF position statement: vitamin D recommendations for older adults. Osteoporos Int. 2010 Jul;21(7):1151-4. doi: 10.1007/s00198-010-1285-3. Epub 2010 Apr 27. PMID 20422154
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Background] Ross AC, Manson JE, Abrams SA, Aloia JF, Brannon PM, Clinton SK, Durazo-Arvizu RA, Gallagher JC, Gallo RL, Jones G, Kovacs CS, Mayne ST, Rosen CJ, Shapses SA. The 2011 Dietary Reference Intakes for Calcium and Vitamin D: what dietetics practitioners need to know. J Am Diet Assoc. 2011 Apr;111(4):524-7. doi: 10.1016/j.jada.2011.01.004. PMID 21443983
- [Background] Heaney RP, Holick MF. Why the IOM recommendations for vitamin D are deficient. J Bone Miner Res. 2011 Mar;26(3):455-7. doi: 10.1002/jbmr.328. PMID 21337617
- [Background] Holick MF, Siris ES, Binkley N, Beard MK, Khan A, Katzer JT, Petruschke RA, Chen E, de Papp AE. Prevalence of Vitamin D inadequacy among postmenopausal North American women receiving osteoporosis therapy. J Clin Endocrinol Metab. 2005 Jun;90(6):3215-24. doi: 10.1210/jc.2004-2364. Epub 2005 Mar 29. PMID 15797954
- [Background] Lyles KW, Colon-Emeric CS, Magaziner JS, Adachi JD, Pieper CF, Mautalen C, Hyldstrup L, Recknor C, Nordsletten L, Moore KA, Lavecchia C, Zhang J, Mesenbrink P, Hodgson PK, Abrams K, Orloff JJ, Horowitz Z, Eriksen EF, Boonen S; HORIZON Recurrent Fracture Trial. Zoledronic acid and clinical fractures and mortality after hip fracture. N Engl J Med. 2007 Nov 1;357(18):1799-809. doi: 10.1056/NEJMoa074941. Epub 2007 Sep 17. PMID 17878149